CLINICAL TRIAL: NCT01580865
Title: Comparison Between Tacrolimus and Mycophenolate Mofetil for Induction of Remission in Lupus Nephritis
Brief Title: Comparison Between Tacrolimus (TAC) and Mycophenolate Mofetil (MMF) for Induction of Remission in Lupus Nephritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other); Maharaj Nakorn Chiang Mai Hospital (Other); Department of Medical Services Ministry of Public Health of Thailand (Other Government); Srinagarind Hospital, Khon Kaen University (Other); Siriraj Hospital (Other); Songklanagarind Hospital (Unknown)
Responsible Party: Principal Investigator, Vasant Sumethkul, Prof., Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRG-LN-11-01
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; Tacrolimus; Mycophenolate mofetil; Complete remission
MeSH Terms: conditions — Lupus Nephritis; Pathologic Complete Response | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Mofetil (MMF) (Active Comparator): MMF was initiated at a dose of 500 mg twice daily (for patients > 50 Kg and Estimated Glomerular Filtration rate (eGFR) > 60 ml/min) for 2 weeks, and advanced to 750 mg twice daily in LN patients weighing less than 50 kg or 1,000 mg twice daily in LN patients weighing 50 kg or more. .
  Interventions: Drug: Tacrolimus vs. Mycophenolate mofetil for Induction Therapy in Lupus Nephritis
- Tacrolimus (TAC) (Experimental): TAC was started at a dosage of 0.1 mg/kg/day divided into 2 daily doses at 12-hour intervals, and the dosage was titrated to achieve trough blood concentrations of 6-10 ng/mL in the first and second month and then 4-8 ng/mL., thereafter
  Interventions: Drug: Tacrolimus vs. Mycophenolate mofetil for Induction Therapy in Lupus Nephritis

INTERVENTIONS:
Drug: Tacrolimus vs. Mycophenolate mofetil for Induction Therapy in Lupus Nephritis — Patients were randomly assigned to receive regimen I or II: TAC plus prednisolone (TAC group) or MMF plus prednisolone (MMF group). TAC was started at a dosage of 0.1 mg/kg/day divided into 2 daily doses at 12-hour intervals, and the dosage was titrated to achieve trough blood concentrations of 6-10 ng/mL in the first and second month and then 4-8 ng/mL., thereafter. MMF was initiated at a dose of 500 mg twice daily (for patients > 50 Kg and Estimated Glomerular Filtration rate (eGFR) > 60 ml/min) for 2 weeks, and advanced to 750 mg twice daily in LN patients weighing less than 50 kg or 1,000 mg twice daily in LN patients weighing 50 kg or more. Patients received concomitant prednisone at a dose of 0.5-0.7 mg/kg/d (maximum 60 mg/day), with tapering by 5-10 mg/day every 2 weeks until a dose of 5 mg/d has been achieved, and this dosage was maintained until the end of 24 weeks.

SUMMARY:
Prospective, multi-center, randomized, controlled, trial to compare tacrolimus with mycophenolate mofetil (MMF) for induces complete remission in lupus nephritis patients. The study duration is one year.

Research hypothesis

* The proportion of patients who have achieved complete remission between regimen of tacrolimus plus prednisolone is greater than MMF plus prednisolone as an induction therapy in lupus nephritis.

DETAILED DESCRIPTION:
The patients with a pathological diagnosis of active lupus nephritis whom are currently followed up or referred to outpatient department (OPD) of 7 participating medical centers in Thailand. Patients who come to attend will be selected according to the inclusion and exclusion criteria.

Outcome measurements

* The patients will be follow-up for 1 year and will be evaluated for clinical manifestations and laboratory investigations of lupus nephritis and any adverse effects of therapy on each visit.
* Blood pressure and laboratory assessments, including complete blood cell count, urinalysis, urine protein creatinine ratio (UPCR), and kidney and liver function, will be performed at each visit for 24 weeks and at the end of study (48 weeks).
* Serum anti-double-stranded DNA antibodies and serum C3 will be measured every 8 weeks after treatment until 24 weeks and at the end of study (48 weeks).
* A fasting lipid profile will be also measured every 8 weeks until 24 weeks and at the end of study (48 weeks).
* Renal and extrarenal disease activity of SLE was measured using the SLEDAI2K. The SLEDAI2K will be evaluated at the time of entry into the study and every 8 weeks after treatment until 24 weeks and at the end of study (48 weeks).
* SLICC damage index, SF-36, EQ5D, and SLEQOL will be evaluated at the time of entry, at 24 weeks, and at the end of the study.
* Patients' serum and urine (blood 3ml and urine 50 ml) will be collected at baseline, 2nd week, 4th week, 12th week, and 48th week for further analysis of biomarkers in the future.

ELIGIBILITY:
Inclusion Criteria:

* The patient who had biopsy-proven lupus nephritis class III, IV or V according to the International Society of Nephrology (ISN)/Renal Pathology Society (RPS) 2003 classification (ISN/RPS2003) within 16 weeks of randomization and had ANA or anti-dsDNA positive.
* Laboratory tests documented the presence of active nephritis, defined as proteinuria (protein excretion >1 g/24 h or spot UPCR > 1 for at least two samples) or increased serum creatinine level (>0.3 mg/dL of baseline but less than 2.0 mg/dl) with active urinary sediment (any of >5 red blood cells/high-power field, >5 white blood cells/high-power field, or red blood cell casts in the absence of infection or other causes).
* Willingness to participate in the study, and be able to read and provide informed consent.

Exclusion Criteria:

* Severe extra-renal manifestations that may require high-dose steroids or other immunomodulating treatments. The definition of severe extra-renal diseases in this investigation are defined by

  * Active central nervous system deemed to be severe or progressive and/ or associated with significant cognitive impairment leading to inability to provide informed consent and/ or comply with the protocol.
  * Any condition, including clinical findings or the laboratory results, which the investigators consider the patients have high disease activity and need high dose steroid and immunosuppressive drugs or other therapy depending on investigator opinion.
  * Severe myocarditis with congestive heart failure or renal failure.
* Previous therapy with calcineurin inhibitor or MMF or CYC within the previous 4 months before randomization.
* Allergy with macrolide antibiotics.
* Uncontrolled hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg) at screening day.
* Severely deteriorated renal function or rapid progressive crescentic Glomerulonephritis.
* Severe myocarditis or cardiomyopathy which may or may not be related to SLE
* Patients who have thrombotic microangiopathy who require treatment with plasmapheresis or IVIG.
* Severe infection or active TB.
* Active hepatitis and evidence of chronic liver disease.
* HIV infection.
* Diabetes mellitus.
* Women who were pregnant or unwilling to use contraception.
* Patients who response to steroid (complete remission) during the run in period (4 weeks).
* Known hypersensitivity or contraindication to MMF, mycophenolic acid (MPA), tacrolimus, corticosteroids or any components of these drug products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Complete remission | 1 year
  Return of serum creatinine to previous baseline, plus a decline in the UPCR to <500 mg/g (<50 mg/mmol)

SECONDARY OUTCOMES:
Partial remission | 1 year
  Stabilization (±25%), or improvement of serum creatinine, but not to normal, plus a ≥50% decrease in UPCR. If there was nephrotic-range proteinuria (UPCR ≥3000 mg/g [≥300 mg/mmol]), improvement requires a ≥50% reduction in UPCR, and a UPCR <3000 mg/g [<300 mg/mmol]
Urine protein to creatinine ratio (UPCR) | 1 year
  g/day
Serum creatinine | 1 year
  mg/dL
Glomerular filtration rate (GFR) | 1 year
  mL/min/1.73m2
Adverse events | 1 year
  Infection, leukopenia, gastrointestinal (GI) symptoms, new onset diabetes mellitus (DM)/hyperglycemia
Serious dverse events | 1 year
  Hospitalization, death
EQ5D | 1 year
  The Euro quality of life -5 Dimensions
SF36 | 1 year
  The 36-Item Short Form Health Survey
SLEQOL | 1 year
  Systemic Lupus Erythematosus Quality of Life Questionnaire
SLEDAI-2K | 1 year
  Systemic Lupus Erythematosus Disease Activity Index 2000

CONTACTS AND LOCATIONS:
Overall Officials: Vasant Sumethkul, Prof., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Ramathibodi Hospital, Rahathevi, Bangkok, Thailand